CLINICAL TRIAL: NCT04801069
Title: Pilot-Study for SAS Treatment in Acute Cerebral InfarctiOn: the PISTACIO Trial
Acronym: PISTACIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SOS Attaque Cérébrale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-A02878-31
Record Dates: First submitted 2021-03-05; First posted 2021-03-16 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Ischemic Stroke; Sleep Apnea Syndromes
MeSH Terms: conditions — Ischemic Stroke; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auto-Adaptative Servo-Ventilation (Experimental)
  Interventions: Device: Nocturnal Ventilation
- Control (No Intervention)

INTERVENTIONS:
Device: Nocturnal Ventilation — AirCurve 10CS PaceWave (Resmed)
  Arms: Auto-Adaptative Servo-Ventilation

SUMMARY:
Sleep Apnea Syndrome (SAS) is highly prevalent in acute stroke and it is related to worst outcome. We aim to assess if SAS treatment, started immediately after acute ischemic stroke, impacts infarct growing and clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke on brain MRI
* NIHSS 6-22
* thrombolysis

Exclusion Criteria:

* Previous SAS
* Previous stroke
* Auto-adaptative Servo-Ventilation Contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Infarct progression | 7 days
  Ischemic size at 7 days compared to ischemic size at admission on brain MRI

SECONDARY OUTCOMES:
Neurological outcome | 3 months
  modified Rankin score (mRS), from 0 (no disability) to 6 (dead)
Neurological outcome on NIHSS | 3 months
  National Institute of Health Stroke Scale (NIHSS), from 0 (normal neurological examination) to 42
Duration of Auto-adaptative Servo-Ventilation use | 7 days
  mean duration per night auto-adaptative servo-ventilation was used during 7 days
SAS prevalence | 3 months
  assessed by respiratory polygraphy
SAS severity | 3 months
  assessed by apnea-hypopnea-index meseared by respiratory polygraphy, mild if AHI is 5-15/h, moderate if AHI is 15-30/h and severe if AHI is > 30/h
Central apnea index | 3 months
  assessed by respiratory polygraphy
Obstructive apnea index | 3 months
  assessed by respiratory polygraphy
Quality of life on SF-12 questionnaire | 3 months
  SF-12 (Short Form Survey 12) questionnaire (not a scale, result is shown as 2 numbers (physical and mental component scores) : if superior to 50, the quality of life is better to the mean quality of life in general population, if less than 50, the quality of life is worse than in the general population)
Quality of sleep on Pittsburgh Sleep Quality Index | 3 months
  Pittsburgh Sleep Quality Index, from 0 (good quality of sleep) to 21 (bas quality of sleep)
Daytime Sleepiness | 3 months
  Epworth Sleepiness Scale, from 0 (no sleepiness) to 24 (great sleepiness), sleepiness if > 10

CONTACTS AND LOCATIONS:
Overall Officials: Elena Meseguer, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Meseguer, Paris, France

IPD SHARING:
Plan to Share IPD: No